CLINICAL TRIAL: NCT03365856
Title: Remission in Rheumatoid Arthritis in the Asian-Pacific Region
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKUPH-R-RA
Record Dates: First submitted 2017-12-04; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RA patients: As routinary clinical practice and observational study
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — as clinical practice

SUMMARY:
This study is the multi-center, open and cross-sectional study of RA remission in Asia Pacific region. The objectives is to explore remission rate of RA patients in different countries in the Asian-Pacific area using different criteria of remission (DAS28, CDAI, SDAI, ACR/EULA remission criteria, RAPID3 and Clin28) and investigate the associated factors of remission in RA patients.

ELIGIBILITY:
Inclusion Criteria:

* RA patients fulfilled the American College of Rheumatology 1987 criteria or the 2010 ACR/EULAR classification criteria.
* Patients aged > 18 years.

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients in our centres are enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
remission rate of RA patients in different countries in the Asian-Pacific area | 12-24 months
  according to the different criteria of clinical remission in RA patients